CLINICAL TRIAL: NCT06010186
Title: Evolution of Muscle Function, Breathlessness and Quality of Life Following Intra or Extra-Abdominal Sepsis in ICU Patients
Acronym: EMBLemAticS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EMBLemAticS
Record Dates: First submitted 2023-08-08; First posted 2023-08-24 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound measurement of the diaphragm and intercostals (Experimental): The specific research procedures correspond to the addition of :
  * Two additional ultrasound examinations, i.e. at discharge from intensive care and 3 months after hospital discharge: non-invasive examination (duration 20 minutes). Ultrasound is a risk-free, painless procedure involving the placement of an ultrasound probe on the body part under investigation, without the need for a radius or puncture.
  * Questionnaires to assess quality of life (SF-36) and functional impact (LCADL) of dyspnea, carried out at discharge from hospital and at 3 months (duration 15 minutes).
  Interventions: Other: Ultrasound measurement of the diaphragm and intercostals

INTERVENTIONS:
Other: Ultrasound measurement of the diaphragm and intercostals — The specific research procedures correspond to the addition of :
  * Two additional ultrasound examinations, i.e. at discharge from intensive care and 3 months after hospital discharge: non-invasive examination (duration 20 minutes). Ultrasound is a risk-free, painless procedure involving the placement of an ultrasound probe on the body part under investigation, without the need for a radius or puncture.
  * Questionnaires to assess quality of life (SF-36) and functional impact (LCADL) of dyspnea, carried out at discharge from hospital and at 3 months (duration 15 minutes).

SUMMARY:
Sepsis is organ dysfunction secondary to an inappropriate host response to infection. In the most severe cases, circulatory failure necessitating the introduction of vasopressor therapy is called septic shock. Sepsis and septic shock are life-threatening systemic organ dysfunctions requiring hospitalization in a critical care unit. According to several studies, sepsis accounts for around 30% of patients in these units. In this patient population, mortality in the critical care unit or in hospital is 25.8% and 35.3% respectively.

Among the organ dysfunctions associated with sepsis, striated skeletal muscle damage is frequent and possibly severe. The literature refers to this as sepsis-induced myopathy, and describes three main mechanisms: mitochondrial dysfunction, exacerbated proteolysis and altered muscle membrane excitability.

Of all the striated skeletal muscles that can be affected, the diaphragm and the muscles of the thoracic and abdominal wall play a major role in breathing. The diaphragm remains the main muscle involved in breathing. Its physiology is twofold. Firstly, through its contraction, the diaphragm is responsible for the lateral movement of the lower ribs, thus increasing the transverse diameter of the thorax. This first action is commonly referred to as "insertional". At the same time, lowering the phrenic center of the diaphragm increases abdominal pressure. Its distinctive upwardly convex domed appearance means that it is intimately in contact with both the chest wall and the abdominal cavity. This particular area of contact is called the apposition zone. It is on this zone, under the action of the abdominal compartment, that positive pressure also generates an outward thrust from the medial face of the lower ribs, a second action commonly referred to as "appositional".

A number of studies, including that carried out by our team (US_DIAMONDS, NCT 02474797), have identified a high prevalence of diaphragmatic damage in patients with sepsis or septic shock. This can be as high as 60%. This diaphragmatic dysfunction would then be associated with a higher mortality rate in hospital and at D90 of discharge.

The clinical evolution of post-resuscitation patients remains a little-studied subject. However, patients may present muscle dysfunctions in the longer term after a stay in intensive care. In our study, we demonstrated that less than half of patients recovered from diaphragmatic dysfunction on discharge from the critical care unit. In addition, Borges RC et al. found a significant decrease in the cross-sectional area of the rectus femoris at discharge, compared with the same measurement taken at D+2 of admission to the critical care unit.

Finally, the impact of muscle dysfunction on dyspnoea during sepsis and after its resolution is uncertain. Similarly, the impact of muscle dysfunction and dyspnoea on quality of life is unknown. Sepsis is associated with muscle dysfunction of multiple mechanisms. The aim of this study is to assess the immediate and longer-term impact of muscle dysfunction on muscle, dyspnea and quality of life in patients with abdominal sepsis ("Abdominal sepsis" group) and patients with extra-abdominal sepsis ("Extra-abdominal" group). Depending on the location of sepsis, this study will enable us to assess and potentially confirm the preferential effect of abdominal sepsis on diaphragm function.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age,
* Patient admitted to a critical care unit at Paris Saint-Joseph Hospital,
* Sepsis or septic shock (defined by the international consensus conference "sepsis-3"),
* Sepsis/septic shock less than 72 hours old,
* Patient affiliated to a health insurance scheme,
* French-speaking patient,
* Patient or relative who has given free, informed and express consent.

Exclusion Criteria:

* History of documented chronic muscular disease, whatever the cause (neuromuscular damage, abdominal or diaphragmatic hernia, muscular damage of inflammatory origin, myopathies, etc.),
* Moribund patients,
* Patient already included in a type 1 interventional research protocol (RIPH1),
* Patient under guardianship,
* Patient deprived of liberty,
* Patient under court protection,
* Pregnant patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2025-07-27 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diaphragm thickening function | Month 3
  This outcome corresponds to the difference in mean ultrasound diaphragm thickening fraction between ICU discharge and 3 months after hospital discharge.

SECONDARY OUTCOMES:
Function of thickening the diaphragm during inspiratory efforts | Month 1
  This outcome corresponds to the difference in mean between the two groups in the fraction of diaphragm thickening, on ultrasound, within the first 72 hours of admission and on discharge from the intensive care unit.
Evolution of diaphragm mobility during inspiratory efforts | Month 3
  This outcome corresponds to the difference in diaphragmatic excursion means within the first 72 hours of admission, at discharge from intensive care and 3 months after hospital discharge.
Evolution of intercostal, transversus abdominis and oblique abdominal muscle function | Month 3
  This outcome corresponds to the comparison of thickness of intercostal, transverse and oblique abdominal muscles within the first 72 hours of admission, on discharge from intensive care and 3 months after hospital discharge.
Evolution of the cross-sectional area of the rectus femoris on ultrasound | Month 3
  This outcome corresponds to the comparison of the cross-sectional area of the rectus femoris within the first 72 hours of admission, on discharge from the intensive care unit and 3 months after hospital discharge.
Evolution of the structure of the various muscle groups assessed by ultrasound | Month 3
  This outcome corresponds to the comparison of gray levels on image captures of different muscle groups using Image J software®.
Global measurement of dyspnea | Month 3
  This outcome corresponds to theVAS-Dyspnea comparison (numerical scale from 0 to 10) within the first 72 hours of admission to intensive care, at discharge from intensive care, at discharge from hospital and 3 months after discharge from hospital.
Functional impact of dyspnea | Month 3
  This outcome corresponds to london chest activity of daily living scale at hospital discharge (estimate of previous condition) and 3 months after discharge. london chest activity of daily living
Short Form-36 Questionnaire of Quality of life | Month 3
  This outcome corresponds to the Short Form-36 comparison at hospital discharge (estimate of previous condition) and 3 months after discharge.
Relationship between diaphragm function and dyspnea, and quality of life | Month 3
  This outcome corresponds to the correlation between diaphragm thickening fraction and LCADL scale, SF-36 quality-of-life questionnaire physical score.

CONTACTS AND LOCATIONS:
Overall Officials: Johan WORMSER, Principal Investigator — Hôpital Paris Saint-Joseph
Locations (1):
- Hôpital Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Demoule A, Jung B, Prodanovic H, Molinari N, Chanques G, Coirault C, Matecki S, Duguet A, Similowski T, Jaber S. Diaphragm dysfunction on admission to the intensive care unit. Prevalence, risk factors, and prognostic impact-a prospective study. Am J Respir Crit Care Med. 2013 Jul 15;188(2):213-9. doi: 10.1164/rccm.201209-1668OC. PMID 23641946
- [Background] Le Neindre A, Wormser J, Luperto M, Bruel C, Misset B, Bouhemad B, Philippart F. Diaphragm function in patients with sepsis and septic shock: A longitudinal ultrasound study. Aust Crit Care. 2023 Mar;36(2):239-246. doi: 10.1016/j.aucc.2022.01.003. Epub 2022 Mar 7. PMID 35272911
- [Background] Vincent JL, Sakr Y, Sprung CL, Ranieri VM, Reinhart K, Gerlach H, Moreno R, Carlet J, Le Gall JR, Payen D; Sepsis Occurrence in Acutely Ill Patients Investigators. Sepsis in European intensive care units: results of the SOAP study. Crit Care Med. 2006 Feb;34(2):344-53. doi: 10.1097/01.ccm.0000194725.48928.3a. PMID 16424713
- [Background] Sakr Y, Jaschinski U, Wittebole X, Szakmany T, Lipman J, Namendys-Silva SA, Martin-Loeches I, Leone M, Lupu MN, Vincent JL; ICON Investigators. Sepsis in Intensive Care Unit Patients: Worldwide Data From the Intensive Care over Nations Audit. Open Forum Infect Dis. 2018 Nov 19;5(12):ofy313. doi: 10.1093/ofid/ofy313. eCollection 2018 Dec. PMID 30555852
- [Background] Hadda V, Kumar R, Tiwari P, Mittal S, Kalaivani M, Madan K, Mohan A, Guleria R. Decline in diaphragm thickness and clinical outcomes among patients with sepsis. Heart Lung. 2021 Mar-Apr;50(2):284-291. doi: 10.1016/j.hrtlng.2020.12.014. Epub 2020 Dec 28. PMID 33383547
- [Background] Borges RC, Soriano FG. Association Between Muscle Wasting and Muscle Strength in Patients Who Developed Severe Sepsis And Septic Shock. Shock. 2019 Mar;51(3):312-320. doi: 10.1097/SHK.0000000000001183. PMID 29757913
- [Background] Bougle A, Rocheteau P, Sharshar T, Chretien F. Muscle regeneration after sepsis. Crit Care. 2016 May 19;20(1):131. doi: 10.1186/s13054-016-1308-3. PMID 27193340
- [Background] De Troyer A, Boriek AM. Mechanics of the respiratory muscles. Compr Physiol. 2011 Jul;1(3):1273-300. doi: 10.1002/cphy.c100009. PMID 23733642
- [Background] Chen Y, Liu Y, Han M, Zhao S, Tan Y, Hao L, Liu W, Zhang W, Song W, Pan M, Jiao G. Quantification of diaphragmatic dynamic dysfunction in septic patients by bedside ultrasound. Sci Rep. 2022 Oct 15;12(1):17336. doi: 10.1038/s41598-022-21702-6. PMID 36243883
- [Background] Laghi FA Jr, Saad M, Shaikh H. Ultrasound and non-ultrasound imaging techniques in the assessment of diaphragmatic dysfunction. BMC Pulm Med. 2021 Mar 15;21(1):85. doi: 10.1186/s12890-021-01441-6. PMID 33722215
- [Background] Solverson KJ, Grant C, Doig CJ. Assessment and predictors of physical functioning post-hospital discharge in survivors of critical illness. Ann Intensive Care. 2016 Dec;6(1):92. doi: 10.1186/s13613-016-0187-8. Epub 2016 Sep 20. PMID 27646108
- [Background] Grassi A, Ferlicca D, Lupieri E, Calcinati S, Francesconi S, Sala V, Ormas V, Chiodaroli E, Abbruzzese C, Curto F, Sanna A, Zambon M, Fumagalli R, Foti G, Bellani G. Assisted mechanical ventilation promotes recovery of diaphragmatic thickness in critically ill patients: a prospective observational study. Crit Care. 2020 Mar 12;24(1):85. doi: 10.1186/s13054-020-2761-6. PMID 32164784
- [Background] Goligher EC, Fan E, Herridge MS, Murray A, Vorona S, Brace D, Rittayamai N, Lanys A, Tomlinson G, Singh JM, Bolz SS, Rubenfeld GD, Kavanagh BP, Brochard LJ, Ferguson ND. Evolution of Diaphragm Thickness during Mechanical Ventilation. Impact of Inspiratory Effort. Am J Respir Crit Care Med. 2015 Nov 1;192(9):1080-8. doi: 10.1164/rccm.201503-0620OC. PMID 26167730
- [Background] Lu Z, Ge H, Xu L, Guo F, Zhang G, Wu Y. Alterations in diaphragmatic function assessed by ultrasonography in mechanically ventilated patients with sepsis. J Clin Ultrasound. 2019 May;47(4):206-211. doi: 10.1002/jcu.22690. Epub 2019 Jan 22. PMID 30671990
- [Background] Le Neindre A, Hansell L, Wormser J, Gomes Lopes A, Diaz Lopez C, Romanet C, Choukroun G, Nguyen M, Philippart F, Guinot PG, Buscher H, Bouhemad B, Ntoumenopoulos G. Thoracic ultrasound influences physiotherapist's clinical decision-making in respiratory management of critical care patients: a multicentre cohort study. Thorax. 2023 Feb;78(2):169-175. doi: 10.1136/thoraxjnl-2021-218217. Epub 2022 Mar 23. PMID 35321941